CLINICAL TRIAL: NCT06394999
Title: Prospective Phase III Multi-center Open-label Study of the Efficacy, Safety, and Acceptability of Mifepristone 50 mg Once-weekly as a Contraceptive
Brief Title: Efficacy, Safety, and Acceptability of Mifepristone 50 mg Once-weekly as a Contraceptive
Acronym: WOMEN&More
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Karolinska Institutet (Other); Women on Waves (Unknown); Children's Investment Fund Foundation (Other)
Responsible Party: Principal Investigator, Rebecca Gomperts, MD, PhD, Researcher, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-502694-41-00
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Female Contraception
Keywords: Oral; Weekly; Non-hormonal
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mifepristone 50 mg (Experimental): mifepristone 50 mg once weekly
  Interventions: Drug: Mifepristone 50 mg

INTERVENTIONS:
Drug: Mifepristone 50 mg — Once-weekly oral mifepristone 50 mg

SUMMARY:
Participants in the study will use mifepristone 50 mg once-a-week for one year as a contraceptive. With this, we want to confirm that the chances of getting pregnant while using this contraceptive are very small. We also want to demonstrate that the use of mifepristone is safe, and it does not lead to any severe health problems. We expect fewer side effects compared to other frequently used contraceptives with hormones. Mifepristone does not contain these hormones. It is important to know how people experience that use of one tablet a week.

DETAILED DESCRIPTION:
Mifepristone 50 mg, a progesterone receptor modulator, is a proven safe emergency contraceptive and a promising new weekly contraceptive. As mifepristone does not contain estrogens or progestogens, we anticipate users will not experience the undesirable side effects and health risks of current hormonal contraceptives. Furthermore, pills are a highly desired formulation approach and a weekly regimen instead of daily administration will likely contribute to a high acceptability and adherence among users. Based on promising early stage clinical data, we expect the use of weekly mifepristone 50 mg as a contraceptive will be safe, effective, and acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35 at the moment of signing the informed consent.
2. In case of 30 years or older, prior HPV or pap-test.
3. Understand and speak Dutch or English.
4. Willing to use mifepristone as the only method of contraception for 12 months.
5. Able to take oral medication and willing to adhere to the study protocol.
6. Have unprotected vaginal heterosexual intercourse with a non-sterilized partner at least once a month.
7. BMI < 35 kg/m2.
8. Willing to fill in a daily diary on the smartphone or computer and five times an on-line questionnaire.
9. Able to participate in the scheduled visits and comply with the study protocol.
10. Provide informed consent about participating in study and provide permission to request medical data in the event of complications or pregnancy.
11. In case of not using hormonal contraceptives, menstrual cycle of 21-35 days.
12. In case of Depo-Provera (3 month injectable) at least 3 cycles of 21-35 days after stop.
13. In case of necessary progesterone treatment, be willing to use condoms temporarily.

Exclusion Criteria:

1. Currently pregnant or breast-feeding.
2. Desire to become pregnant within the following 12 months.
3. Signs of current endometritis, incomplete abortion after miscarriage or induced abortion, or retained pla-cental rests after delivery.
4. Undiagnosed post-coital bleeding or unscheduled bleeding (spotting with COC, patch, vaginal ring, hormo-nal IUD, implant allowed).
5. Known subfertility or history of ectopic pregnancy, unless intra-uterine pregnancy afterwards, or grade 3-4 endometriosis proven by laparoscopy.
6. History of gastric reduction or gastric bypass or use of weight-loss medicines.
7. Previous or current liver illness, previous or current infection affecting the liver (such as Hepatitis) or mod-erately abnormal liver enzymes at screening (ALAT, ASAT or bilirubin > 2 ULN).
8. Current or previous cancer or DCIS.
9. Family history of endometrial cancer, except BRCA genome mutation.
10. Known allergy to mifepristone.
11. Using non-dermal corticosteroids or any drugs that may interact with mifepristone. These include hydan-toins (e.g. phenytoin), barbiturates (e.g. phenobarbital), primidone, carbamazepine, rifampicin, oxcarbaze-pine, topiramate, rifabutin, felbamate, ritonavir, nelfinavir, griseofulvin and products containing St. John's wort (Hypericum perforatum).
12. Treatment with another investigational drug or participating in another intervention study, unless the prin-cipal investigators agree.
13. Undiagnosed reason for severe anemia or increased creatinine.
14. Abnormal previous PAP smear > pap II without colposcopic evaluation or untreated HSIL.
15. Systolic blood pressure ≥ 180 mmHg and/or diastolic ≥ 110 mmHg (hypertension with medical treatment allowed).
16. Intracavitary abnormalities on vaginal ultrasound, including intracavitary polyps or myomas, endometrium > 15 mm, or an obvious sign of hydrosalpinx.
17. Previous participation in the WOMEN&More trial.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1186 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Overall Pearl Index | 0-12 months
  Nominator Number of pregnancies with conception during treatment period from the first day of pill intake to the last day of pill intake + 7 days
  Denominator The time period from the first day of pill intake to the last day of pill intake + 7 days. Cycles with documentation of no unprotected intercourse will be subtracted from this period, unless in the unlikely case that a pregnancy occurred in such a cycle.
Pearl Index by Method failure | 0-12 months
  Nominator Number of pregnancies with conception during cycles as defined in the denominator
  Denominator The number of cycles with perfect use times 1300. A cycle is defined as (at least) 28 days after the first day of mifepristone 50 mg intake. Cycles with documentation of no unprotected intercourse will be subtracted from this time period, unless in the unlikely case that a pregnancy occurred in such a cycle. Also, cycles with non-perfect use, i.e. without mifepristone 50 mg intake at least once every 7 days will be excluded. Diary charts and counting of remaining tablets will provide dosing information to determine (non-) perfect use.
Assess the contraceptive safety of once-weekly mifepristone 50 mg | 3, 6 and 12 months
  Proportion of women with endometrial thickness >15 mm, endometrium with irregular cystic appearance on US; with ALT, AST elevation three times above normal levels or bilirubin two times above normal levels; with adverse events / serious adverse events

SECONDARY OUTCOMES:
Depression | baseline, 3, 6 and 12 months
  PHQ-9 questionnaire (mean value) and changes
Sexual functioning | baseline, 3, 6 and 12 months
  Female Sexual Function Index (FSFI) (mean value) and changes
Use of antidepressants | baseline, 3, 6 and 12 months
  Proportion of participants who use antidepressants or mood stabilizing drugs
Weight [kg] | baseline, 3, 6 and 12 months
  Weight changes
Bleeding profile | 0-365 days
  Daily reported bleeding pattern and changes in bleeding pattern regarding amount of bleeding, pain, use of painkillers and effect on hemoglobin
Side effects | 0-365 days
  Proportion of participants with daily reported side-effects and changes
Acceptability | 3, 6 and 12 months
  Proportion of participants who find the medication acceptable
Liver function | 3, 6 and 12 months
  Frequency of abnormal liver functions between 2 and 3 x ULN (ALT/AST) and time to become less than 2 x ULN
Pregnancy outcomes | 21 months
  Number of abortions, miscarriages, ectopic pregnancies, preterm labor, growth restriction and congenital abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gomperts, PhD, Principal Investigator — Leiden University Medical Center
Locations (14):
- Netherlands (14):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Flevoziekenhuis, Almere Stad
  - Amsterdam Universitair Medische Centra, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Admiraal De Ruyter Ziekenhuis, Goes
  - Martini Ziekenhuis, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Franciscus Gasthuis, Rotterdam
  - Diakonessenhuis, Utrecht
  - Maxima Medisch Centrum, Veldhoven